CLINICAL TRIAL: NCT02176993
Title: Effects of Surface Cooling On Stroke Outcome triaL: a Feasibility and Safety Study
Brief Title: Effects of Surface Cooling On Stroke Outcome triaL (COOL)
Acronym: COOL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Robbert-Jan van Hooff, M.D., Ph.D., Universitair Ziekenhuis Brussel
Other Study IDs: B.U.N. 143201215226
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Acute Stroke; Hypothermia
Keywords: Acute stroke; Therapeutic Hypothermia
MeSH Terms: conditions — Stroke; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Application of surface cooling: Surface cooling during 60 minutes.

SUMMARY:
The investigators goal is to improve the outcome of patients with acute stroke by inducing mild cerebral hypothermia through surface cooling at the cervical and shoulder regions using EMCOOLS Brain.Pads®.

For this project, the investigators can build further on their research group's experience with hypothermia in animal models and invasive cooling in stroke patients.

The COOL program will prospectively evaluate safety, feasibility, patient acceptance and efficacy of mild cerebral hypothermia using EMCOOLS Brain.Pads® in a large cohort of patients presenting with acute stroke at the Emergency Department of the Universitair Ziekenhuis Brussel. The application of EMCOOLS Brain.Pads® will be compared to routine clinical practice in a randomized controlled trial. If proven to be safe, feasible, well-tolerated and efficacious in the inhospital setting, future use in prehospital acute stroke care will be incorporated with telemedicine support, as part of the Prehospital Stroke Study at the Universitair ziekenhuis Brussel (PreSSUB).

DETAILED DESCRIPTION:
Several studies have identified fever as an independent predictor of poor outcome in patients with acute stroke. Experimental data and clinical studies indicate that therapeutic hypothermia has neuroprotective effects associated with better clinical outcome, probably through reduction of infarct volume and cerebral edema in patients with ischemic and hemorrhagic stroke, respectively. It is to be expected that the beneficiary effects of hypothermia will be more pronounced if initiated early after stroke onset, which underlines the rational that this technique ideally should be initiated in the prehospital phase of acute stroke management.

Therapeutic hypothermia can be obtained by external or by endovascular cooling. Most methods aim to lower the body temperature to <33°C and therefore require patient sedation and intubation. In contrast to patients with cardiac arrest, sedation and intubation preferably are avoided and profound cooling of the entire body is not desired nor required in in stroke patients. EMCOOLS pads® have originally been developed by EMCOOLS Medical Cooling Systems AG (Austria) for profound external cooling of patients with cardiac arrest. The novel EMCOOLS Brain.Pad® was redesigned to mildly lower the brain temperature through noninvasive surface cooling of the cerebropetal arteries at the cervical level. Pilot studies in healthy volunteers demonstrated that a decrease of 0.5-1°C (tympanic measurement) can be safely obtained by application of EMCOOLS Brain.Pad® during 60 to 90 minutes. No relevant side effects were observed in these small studies, but possible effects on cerebrovascular blood flow were not evaluated.

Early application of mild therapeutic hypothermia in acute stroke patients builds further on their research group's experience with hypothermia in animal models and stroke patients. The investigators propose a prospective clinical trial comparing current clinical practice with the induction of mild hypothermia using EMCOOLS Brain.Pads® in patients presenting with acute stroke. If safety, feasibility, patient acceptance and efficacy are confirmed in the inhospital setting, the next step will involve evaluation of this approach in prehospital acute stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Acute stroke with onset < 24 hours

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient older than 18 year presenting with an acute stroke and onset < 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of neurological deficit as measured by NIHSS | 90 days post-stroke
  The National Institute of Health Stroke Scale (NIHSS) will be used as a measure to assess the gain in neurological deficit 90 days post-stroke.

SECONDARY OUTCOMES:
Temperature change during surface cooling | During cooling and 30 minutes thereafter
  Changes in temperature will be measured with mastoid, inguinal, tympanic and temporal thermometers.

OTHER OUTCOMES:
Long-term functional outcome | 3 months post-stroke
  The functional outcome will be measured by the modified Rankin Scale (mRS).
Mortality rate | 3 months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Robbert-Jan van Hooff, M.D., Ph.D., Principal Investigator — Universitair Ziekenhuis Brussel Belgium
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium